CLINICAL TRIAL: NCT02446717
Title: A Randomized, Open-Label, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Co-Administration of ABT-493 and ABT-530 (or ABT-493/ABT-530) With and Without Ribavirin in Adults With Chronic Hepatitis C Virus (HCV) Infection Who Failed a Prior Direct-Acting Antiviral Agent (DAA)-Containing Therapy
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of ABT-493 and ABT-530 With and Without Ribavirin in Adults With HCV Who Failed a Prior DAA Containing Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-410; 2015-002350-13 (EudraCT Number)
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Chronic Hepatitis C; Hepatitis C Virus; HCV; Direct-Acting Antiviral Agent (DAA)-Experienced
Keywords: Hepatitis C; HCV Genotype 6; HCV GT1; Interferon (IFN) free; HCV Genotype 5; HCV; HCV GT4; HCV Genotype 4; Chronic Hepatitis C; Chronic HCV; Hepatitis C Genotype 1; HCV GT5; HCV Genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — glecaprevir; pibrentasvir; ombitasvir; glecaprevir and pibrentasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm A (Experimental): ABT-493 (200 mg) once daily (QD) co-administered with ABT-530 (80 mg) QD for 12 weeks in chronic HCV genotype 1- infected participants without cirrhosis.
  Interventions: Drug: ABT-493, ABT-530
- Arm B (Experimental): ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD plus ribavirin (RBV) for 12 weeks in chronic HCV genotype 1- infected participants without cirrhosis.
  Interventions: Drug: ABT-493, ABT-530; Drug: ribavirin (RBV)
- Arm C (Experimental): ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 12 weeks in chronic HCV genotype 1- infected participants without cirrhosis.
  Interventions: Drug: ABT-493, ABT-530
- Arm D (Experimental): ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 12 weeks in HCV genotypes 1- or 4-6- infected participants with or without cirrhosis.
  Interventions: Drug: ABT-493/ABT-530
- Arm E (Experimental): ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 16 weeks in HCV genotype 1- or 4-6- infected participants with or without cirrhosis.
  Interventions: Drug: ABT-493/ABT-530

INTERVENTIONS:
Drug: ABT-493, ABT-530 — ABT-493 (tablet) dosed with ABT-530 (tablet)
  Other Names: ABT-493 also known as glecaprevir; ABT-530 also known as pibrentasvir; ABT-493/ABT-530 (ABT-493 coformulated with ABT-267) also known as MAVYRET
  Arms: Arm A; Arm B; Arm C
Drug: ribavirin (RBV) — Tablet
  Arms: Arm B
Drug: ABT-493/ABT-530 — Tablet; ABT-493 coformulated with ABT-530
  Other Names: ABT-493 also known as glecaprevir; ABT-530 also known as pibrentasvir; MAVYRET
  Arms: Arm D; Arm E

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ABT-493 and ABT-530 with or without ribavirin (RBV) in participants with chronic hepatitis C virus, (HCV)-infection who previously failed treatment with a direct acting antiviral (DAA)-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from 18 to 70 years in Arms A, B, and C; patients 18 years of age or older in Arms D and E.
2. Previous treatment with DAA-containing regimen for chronic hepatitis C virus (HCV) infection resulting in either on-treatment virologic failure or post-treatment relapse
3. Chronic HCV genotype (GT) 1, 4, 5, or 6-infection (GT4-6 in Arms D and E)

Exclusion Criteria:

1. History of severe, life-threatening or other significant sensitivity to any drug
2. Female who is pregnant, planning to become pregnant during the study or breastfeeding; or male whose partner is pregnant or planning to become pregnant during the study
3. Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol
4. Positive for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab)
5. Co-infection with more than one HCV genotype

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Result] Poordad F, Felizarta F, Asatryan A, Sulkowski MS, Reindollar RW, Landis CS, Gordon SC, Flamm SL, Fried MW, Bernstein DE, Lin CW, Liu R, Lovell SS, Ng TI, Kort J, Mensa FJ. Glecaprevir and pibrentasvir for 12 weeks for hepatitis C virus genotype 1 infection and prior direct-acting antiviral treatment. Hepatology. 2017 Aug;66(2):389-397. doi: 10.1002/hep.29081. Epub 2017 Apr 10. PMID 28128852
- [Derived] Brown A, Welzel TM, Conway B, Negro F, Brau N, Grebely J, Puoti M, Aghemo A, Kleine H, Pugatch D, Mensa FJ, Chen YJ, Lei Y, Lawitz E, Asselah T. Adherence to pan-genotypic glecaprevir/pibrentasvir and efficacy in HCV-infected patients: A pooled analysis of clinical trials. Liver Int. 2020 Apr;40(4):778-786. doi: 10.1111/liv.14266. Epub 2019 Oct 18. PMID 31568620
- [Derived] Back D, Belperio P, Bondin M, Negro F, Talal AH, Park C, Zhang Z, Pinsky B, Crown E, Mensa FJ, Marra F. Efficacy and safety of glecaprevir/pibrentasvir in patients with chronic HCV infection and psychiatric disorders: An integrated analysis. J Viral Hepat. 2019 Aug;26(8):951-960. doi: 10.1111/jvh.13110. Epub 2019 May 20. PMID 30977945
- [Derived] Gane E, Poordad F, Zadeikis N, Valdes J, Lin CW, Liu W, Asatryan A, Wang S, Stedman C, Greenbloom S, Nguyen T, Elkhashab M, Worns MA, Tran A, Mulkay JP, Setze C, Yu Y, Pilot-Matias T, Porcalla A, Mensa FJ. Safety and Pharmacokinetics of Glecaprevir/Pibrentasvir in Adults With Chronic Genotype 1-6 Hepatitis C Virus Infections and Compensated Liver Disease. Clin Infect Dis. 2019 Oct 30;69(10):1657-1664. doi: 10.1093/cid/ciz022. PMID 30923816
- [Derived] Flamm S, Reddy KR, Zadeikis N, Hassanein T, Bacon BR, Maieron A, Zeuzem S, Bourliere M, Calleja JL, Kosloski MP, Oberoi RK, Lin CW, Yu Y, Lovell S, Semizarov D, Mensa FJ. Efficacy and Pharmacokinetics of Glecaprevir and Pibrentasvir With Concurrent Use of Acid-Reducing Agents in Patients With Chronic HCV Infection. Clin Gastroenterol Hepatol. 2019 Feb;17(3):527-535.e6. doi: 10.1016/j.cgh.2018.07.003. Epub 2018 Sep 10. PMID 30012435
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 42-day screening period.
Period: Overall Study
Arm/Group | ARM A | ARM B | ARM C | ARM D | ARM E
Started | 6 | 22 | 22 | 44 | 47
Completed | 6 | 21 | 20 | 43 | 46
Not Completed | 0 | 1 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 1
Not completed — Withdrew consent | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM A | ARM B | ARM C | ARM D | ARM E | Total
Number analyzed (Participants) | 6 | 22 | 22 | 44 | 47 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (9.16) | 55.2 (6.29) | 58.5 (6.56) | 55.6 (8.57) | 55.6 (8.31) | 55.9 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 13 | 14 | 36
  Male | 3 | 20 | 18 | 31 | 33 | 105

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat population: all participants who received at least 1 dose of study drug; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ARM A | ARM B | ARM C | ARM D | ARM E
Number analyzed (Participants) | 6 | 22 | 22 | 44 | 47
percentage of participants | 100 [61.0 to 100.0] | 95.5 [78.2 to 99.2] | 86.4 [66.7 to 95.3] | 88.6 [76.0 to 95.0] | 91.5 [80.1 to 96.6]

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks Post-treatment (SVR4)
Description: SVR4 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 4 weeks after the last dose of study drug.
Time Frame: 4 weeks after the last actual dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population); participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ARM A | ARM B | ARM C | ARM D | ARM E
Number analyzed (Participants) | 6 | 22 | 22 | 44 | 47
percentage of participants | 100.0 [61.0 to 100.0] | 95.5 [78.2 to 99.2] | 95.5 [78.2 to 99.2] | 90.9 [78.8 to 96.4] | 91.5 [80.1 to 96.6]

3. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ 100 IU after HCV RNA < LLOQ during treatment; confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment; or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: Day 3, Treatment Weeks 1, 2, 4, 6, 8, 10, 12 (end of treatment for 12-week treatment arms), and 16 (end of treatment for 16-week treatment arm) or premature discontinuation from treatment
Population: All participants who received at least 1 dose of study drug (ITT population)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ARM A | ARM B | ARM C | ARM D | ARM E
Number analyzed (Participants) | 6 | 22 | 22 | 44 | 47
percentage of participants | 0.0 [0.0 to 39.0] | 0.0 [0.0 to 14.9] | 4.5 [0.8 to 21.8] | 2.3 [0.4 to 11.8] | 8.5 [3.4 to 19.9]

4. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants with HCV RNA levels < LLOQ at the end of treatment, excluding reinfection.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ARM A | ARM B | ARM C | ARM D | ARM E
Number analyzed (Participants) | 6 | 21 | 21 | 43 | 43
percentage of participants | 0.0 [0.0 to 39.0] | 4.8 [0.8 to 22.7] | 0.0 [0.0 to 15.5] | 9.3 [3.7 to 21.6] | 0.0 [0.0 to 8.2]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 20 weeks).
Description: TEAEs and TESAEs are defined as any AE or SAE with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | ARM A | ARM B | ARM C | ARM D | ARM E
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/22 | 0/22 | 1/44 | 2/47
Other Adverse Events (participants affected / at risk) | 4/6 | 17/22 | 16/22 | 23/44 | 27/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARM A (N=6) | ARM B (N=22) | ARM C (N=22) | ARM D (N=44) | ARM E (N=47)
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
WOUND INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARM A (N=6) | ARM B (N=22) | ARM C (N=22) | ARM D (N=44) | ARM E (N=47)
DRY EYE (Eye disorders) | 1 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 4
DIARRHOEA (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 2
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 4
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 6 | 3 | 4 | 3
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
ASTHENIA (General disorders) | 0 | 0 | 1 | 1 | 3
FATIGUE (General disorders) | 1 | 8 | 4 | 3 | 5
NASOPHARYNGITIS (Infections and infestations) | 0 | 3 | 1 | 1 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1 | 1 | 4
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1 | 2
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 5 | 8 | 6 | 11
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
LETHARGY (Nervous system disorders) | 0 | 0 | 0 | 3 | 1
SOMNOLENCE (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 1 | 2 | 0 | 2
INSOMNIA (Psychiatric disorders) | 0 | 6 | 0 | 2 | 2
IRRITABILITY (Psychiatric disorders) | 0 | 2 | 0 | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.